CLINICAL TRIAL: NCT06757725
Title: Renal Resistive Index as an Indicator of Lupus Nephritis Severity and Systemic Lupus Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Tarek Samy Abdelaziz, Associate professor of Internal medicine and nephrology, Kasr El Aini Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MS-632-2022; MS-632-2022 (Other: Cairo University hospitals)
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Systemic Lupus Erthematosus; Lupus Glomerulonephritis; Lupus Flare
Keywords: systimc lupus erythromatosus; lupus glomerulonephritis
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with lupus nephritis (Active Comparator): Theses are 25 patients diagnosed with lupus nephritis
  Interventions: Diagnostic Test: colour doppler of the renal artery and measurement of resistive index
- Lupus without nephritis (Active Comparator): Theses are 25 patients diagnosed with lupus without evidence of nephritis
  Interventions: Diagnostic Test: colour doppler of the renal artery and measurement of resistive index
- Healthy control (No Intervention): Patients who are healthy volunteers with no evidence of nephritis or systemic lupus

INTERVENTIONS:
Diagnostic Test: colour doppler of the renal artery and measurement of resistive index — using colour doppler to asses vascular resistance and resistive index
  Arms: Lupus without nephritis; Patients with lupus nephritis

SUMMARY:
The study explores the role of the colour Doppler scanning of the renal arteries and its relation to the degree of disease affection in lupus nephritis

DETAILED DESCRIPTION:
we have recruited patients into 3 groups The first group is patients with lupus nephritis The second groups is patients with systemic lupus erythromatosus without nephritis The third groups is normal healthy controls we explored the association of colour Doppler and the renal resistive index with the degree of the renal affection in lupus nephritis

ELIGIBILITY:
Inclusion Criteria:

* 1. Systemic lupus erythematosus. 2. Lupus nephritis. 3. Adults >18 years old.

Exclusion Criteria:

* 1. End Stage Renal Disease. 2. Diabetes Mellitus. 3. Heart failure. 4. Hepatic diseases. 5. Obstructive nephropathy. 6. Renal artery stenosis or occlusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-09-03 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Resistive index | At the time of recruitment
  The resistive index of the renal arteries as measured by the colour Doppler

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Can be shared upon reasonable request